CLINICAL TRIAL: NCT01908387
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study of Oral Azacitidine (CC-486) in Japanese Subjects With Hematological Neoplasms
Brief Title: Phase 1 Study of CC-486 in Japanese Subjects With Hematological Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to Slow Accrual study was terminated.
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-MDS-001
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia; Multiple Myeloma; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Oral azacitidine; CC-486; Hematological neoplasms; Phase 1
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Hematologic Neoplasms | interventions — Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral azacitidine (Experimental)
  Interventions: Drug: Oral azacitidine

INTERVENTIONS:
Drug: Oral azacitidine — 100 mg to 300 mg oral azacitidine once daily for 14 days or 21 days of the initial 28-day cycle
  Other Names: CC-486

SUMMARY:
To identify the maximum tolerated dose (MTD) of oral azacitidine on different treatment schedules in Japanese subjects with hematological neoplasms

DETAILED DESCRIPTION:
This is a phase 1, multicenter, open-label, dose-escalation study that will evaluate the maximum tolerated dose (MTD), safety, pharmacokinetics, and preliminary efficacy of CC-486 in Japanese subjects with hematological neoplasms including myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMML), acute myeloid leukemia (AML), multiple myeloma (MM), non-Hodgkin lymphoma (NHL), or Hodgkin lymphoma (HL). A standard phase 1 design for MTD determination, an open label, dose ascending, "3 + 3" design, is adopted in this study. This study consists of screening phase, MTD determination phase, and treatment phase. Each subject continues study treatment until documentation of progressive disease or discontinuation of study treatment for any reason. Originally only MDS subjects were targeted and the MTD of CC-486 when administered once daily (QD) for 21 days in a 28-day cycle would be evaluated in this study. Currently CC-486 is being clinically developed with both 14-day and 21-day dosing schedules in various diseases. This study was suspended to amend protocol to evaluate the MTD on these different dosing schedule in larger population. This study was re-opened after amended protocol was approved by institutional review board at study site.

ELIGIBILITY:
Inclusion Criteria:

* 1. Eighteen years of age to 80 years of age at the time of signing the informed consent document; 2. Understand and voluntarily sign an informed consent document prior to any study related assessments and/or procedures being conducted; 3. Able to adhere to the study visit schedule and other protocol requirements; 4. Have a documented diagnosis of one of the following:

  * Myelodysplastic syndromes or Chronic myelomonocytic leukemia (based on a bone marrow aspirate or bone marrow biopsy) or;
  * Acute myeloid leukemia (based on a bone marrow aspirate or bone marrow biopsy), limited to those subjects for whom standard curative or palliative measures do not exist or are no longer effective or;
  * Multiple myeloma, limited to those subjects for whom standard curative or palliative measures do not exist or are no longer effective or;
  * Non-Hodgkin lymphoma or Hodgkin lymphoma, limited to those subjects for whom standard curative or palliative measures do not exist or are no longer effective; 5. For subjects with myelodysplastic syndromes only, have at least one of the following:
  * Hemoglobin level ≤ 9.0 g/dL;
  * Platelet count ≤ 75,000 /μL;
  * Red blood cell transfusion-dependent as defined by:
* Average red blood cell transfusion requirement of ≥ 4 units per 28 days confirmed for a minimum of 84 days prior to starting study treatment. Hemoglobin levels within 7 days prior to administration of an red blood cell transfusion must be ≤ 9.0 g/dL in order for the transfusion to be counted towards red blood cell transfusion-dependent status. Red blood cell transfusions administered when hemoglobin levels were > 9.0 g/dL and/or red blood cell transfusions administered for elective surgery will not qualify as a required transfusion for the purpose of providing evidence of red blood cell transfusion-dependent status. Note that 4 units of red blood cell in Japan is equivalent to 2 units of red blood cell outside of Japan;
* No consecutive 42 days that are red blood cell -transfusion-free during the 84 days prior to starting study treatment;

  • Platelet transfusion-dependent as defined by:
* Have at least two separate platelet transfusion episodes during 56 days prior to starting study treatment. Platelet transfusions administered for elective surgery will not qualify as a required transfusion for the purpose of providing evidence of platelet transfusion-dependent status;
* No consecutive 28 days that are platelet-transfusion-free during the 56 days prior to starting study treatment; 6. Eastern Cooperative Oncology Group performance status of 0 or 1; 7. Females of childbearing potential (FCBP: a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal [ie, amenorrhea following cancer therapy does not rule out childbearing potential] for at least 24 consecutive months [ie, has had menses at any time in the preceding 24 consecutive months]) must:

  * Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner; injectable and implantable hormonal contraceptive have not been approved in Japan as of March 2013) throughout the study, and for 3 months following the last dose of oral azacitidine and;
  * Have a negative serum pregnancy test (sensitivity of at least 25 mIU/mL) at screening and;
  * Have a negative urine pregnancy test within 72 hours prior to starting study treatment (note that the screening serum pregnancy test can be used as the test prior to starting study treatment if it is performed within the 72 hour timeframe); 8. Male subjects with a female partner of childbearing potential must agree to use at least 2 physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last dose of study drug.

Exclusion Criteria:

1. Hypoplastic myelodysplastic syndromes defined as bone marrow cellularity of < 20%;
2. Atypical chronic myeloid leukemia and unclassifiable myeloproliferative neoplasms. Subjects with white blood cell counts ≥ 12,000/μL must be excluded (for subjects with acute myeloid leukemia: subjects with white blood cell counts ≥ 15,000/μL must be excluded, and for subjects with chronic myelomonocytic leukemia: subjects with white blood cell counts ≥ 20,000/μL must be excluded);
3. Active central nerve system lymphoma unless the subject has been previously treated and remains asymptomatic for 3 months;
4. Dry tap bone marrow aspirate due to myelofibrosis, and/or myelofibrosis accompanied by splenomegaly;
5. Percentage of neoplasm cells in bone marrow more than 50%;
6. Prior treatment with azacitidine or other hypomethylating agent that was discontinued due to adverse event related to that therapy except adverse events related to topical reactions related to injection of azacitidine;
7. Prior allogeneic or autologous stem cell transplant;
8. History of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity;
9. Thrombocytopenia secondary to other possible causes, including medication(s), congenital disorder(s), immune disorder(s) (eg, idiopathic thrombocytopenic purpura [ITP]), or microvascular disorder(s) (eg, disseminated intravascular coagulation, hemolytic uremic syndrome, thrombotic thrombocytopenic purpura);
10. Treatment with any anticancer therapy (standard or investigational) within the previous 21 days prior to the first dose of study drug or less than full recovery (CTCAE grade 1) from the clinically significant toxic effects of that treatment. Treatment with hydroxyurea within the previous 28 days prior to the first dose of study drug must be excluded;
11. Concurrent use of corticosteroids, except for subjects on a stable or decreasing dose for at least 1 week prior to starting study treatment for medical conditions other than primary diseases. Topical use of corticosteroids is permitted regardless of dose
12. Prior history of malignancies, other than myelodysplastic syndromes, chronic myelomonocytic leukemia, acute myeloid leukemia, multiple myeloma, non-hodgkin lymphoma, or hodgkin lymphoma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following:

    * Basal or squamous cell carcinoma of the skin;
    * Carcinoma in situ of the cervix or breast;
    * Incidental histological finding of prostate cancer (Tumor nodes metastasis [TNM] stage of T1a N0M0 or T1b N0M0);
    * Early-stage gastric cancer suitable for endoscopic mucosal resection or endoscopic submucosal dissection;
13. Significant active cardiac disease within the previous 6 months, including:

    * New York Heart Association (NYHA) class III-IV congestive heart failure;
    * Unstable angina or angina requiring surgical or medical intervention;
    * Myocardial infarction;
14. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment);
15. Known human immunodeficiency virus (HIV) positivity (eg, subjects who are receiving antiretroviral therapy for HIV disease);
16. Hepatitis Bs (HBs) antigen-positive, or hepatitis C virus (HCV) antibody-positive. In case HBc antibody and/or HBs antibody is positive even if HBs antigen-negative, a hepatitis B virus (HBV) DNA test should be performed and if positive the subject will be excluded;
17. Any of the following laboratory abnormalities:

    * Absolute neutrophil count < 1,000/μL (except for subjects with acute myeloid leukemia);
    * Serum glutamic oxaloacetic transaminase/aspartate transaminase or serum glutamic pyruvate transaminase/alanine transaminase > 2.5 ×upper limit of normal;
    * Serum bilirubin > 1.5 × upper limit of normal. High levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis). Subjects are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Coombs' test or over 50% of indirect bilirubin;
    * Serum creatinine > 1.5 × upper limit of normal;
    * Bicarbonate (venous blood) < 22 mEq/L;
    * Abnormal coagulation parameters (Prothrombin time-international normalized ratio > 1.5 or activated partial thromboplastin time > 40 seconds);
    * Hemoglobin level < 8.0 g/dL (for multiple myeloma, non-hodgkin lymphoma, or hodgkin lymphoma only);
    * Platelet count < 25,000 /μL (for multiple myeloma, non-hodgkin lymphoma, or hodgkin lymphoma only);
18. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding;
19. History of cerebrovascular accident or transient cerebral ischemic attack within 6 months prior to starting study treatment;
20. Interstitial lung disease, pulmonary fibrosis, or other severe respiratory disease;
21. Hepatic cirrhosis, or other moderate to severe hepatic disease;
22. Known or suspected hypersensitivity to azacitidine or mannitol;
23. Pregnant or breastfeeding females;
24. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study;
25. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study;
26. Any condition that confounds the ability to interpret data from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | For 28 days
  Number of subjects experiencing dose limiting toxicity during the first 28-day cycle

SECONDARY OUTCOMES:
Number of participants with adverse events. | Up to 4 years
  Number of participants with adverse events. An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria below), regardless of etiology.
Pharmacokinetics - Cmax | On day 1 and day 8
  Maximum observed concentration in plasma
Pharmacokinetics - Tmax | On day 1 and day 8
  Observed time to first maximum plasma concentration
Pharmacokinetics - AUCt | On day 1 and day 8
  Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear trapezoidal rule
Pharmacokinetics - AUC Zero to Infinity | On day 1 and day 8
  Area under the plasma concentration-time curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity will be calculated according to the following equation: AUC∞ = AUCt + (Ct/λz), where Ct is the last quantifiable concentration If the percentage of AUC extrapolated is ≥ 25%, AUC∞ will not be reported.
Pharmacokinetics - AUCext% | On day 1 and day 8
  Percentage of AUC∞ due to extrapolation from the time from the last quantifiable concentration to infinity, calculated as (AUC∞ - AUCt) / AUC∞ ×100
Pharmacokinetics - Terminal Phase | On day 1 and day 8
  Terminal phase rate constant, determined by linear regression of the terminal points of the log-linear plasma concentration-time curve Visual assessment may be used to identify the terminal linear phase of the concentration versus time profile. A minimum of three data points will be used for calculation. λz will not be estimated if the terminal phase of the log-concentration versus time profile does not exhibit a linear decline phase, or if the regression coefficient < 0.8.
Pharmacokinetics - Terminal Half-Life | On day 1 and day 8
  Terminal phase half-life, will be calculated according to the following equation: t1/2 = 0.693/λz
Pharmacokinetics - Total Clearance | On day 1 and day 8
  Apparent total clearance, calculated as Dose/AUC∞
Pharmacokinetics - Volume of distribution | On day 1 and day 8
  Apparent volume of distribution will be calculated according to the equation: Vz/F = (CL/F)/λz
Pharmacokinetics - Aet | On day 1 and day 8
  Cumulative amount excreted from time zero to time t (ng), calculated as the summation of the amounts (Aet, product of urine volume and urine concentration) excreted in subsequent collection intervals
Pharmacokinetics - fet | On day 1 and day 8
  Cumulative fraction of dose excreted in the urine from time zero to time t (%), calculated as Ae t divided by dose
Pharmacokinetics - Renal Clearance | On day 1 and day 8
  Renal clearance (mL/min), calculated as Aet divided by AUCt
Investigator's response assessment | Up to 4 years
  Number of participants who demonstrate response by investigator's assessment based on International Working Group (IWG) criteria Myelodysplastic Syndrome (MDS), Chronic myelomonocytic Leukemia (CMML) and Acute Myeloid (AML), IMWG criteria for Multiple Myeloma (MM), and modified Cheson 2007 criteria for Non-Hodgkin's Lymphoma (NHL) or Hodgkin's Lymphoma (HL)

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Director, Study Director — Celgene K.K.
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Tokyo, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo, Tokyo